CLINICAL TRIAL: NCT01104935
Title: Evaluation of Trastuzumab Without Chemotherapy as a Postoperative Adjuvant Therapy in HER2 Positive Elderly Breast Cancer Patients: Randomized Controlled Trial
Brief Title: National Surgical Adjuvant Study of Breast Cancer(N-SAS BC) 07 [RESPECT]
Acronym: RESPECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Comprehensive Support Project for Oncology Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-SAS BC 07
Record Dates: First submitted 2009-11-06; First posted 2010-04-16 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Drug Therapy; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trastuzumab monotherapy (Experimental): H group (trastuzumab monotherapy group)
  * Trastuzumab: 1-year treatment
  * Loading dose, 8 mg/kg; from 2nd dose, 6 mg/kg; iv inj, qw, 18 times
  Interventions: Drug: trastuzumab monotherapy
- trastuzumab and chemotherapy (Active Comparator): H+CT group (combination therapy of trastuzumab and chemotherapy)
  * Chemotherapy: 12 to 24 weeks
  * Select chemotherapy from certain regimens (PTX, DTX, TC, AC, EC, FEC, CMF and TCb (CBDCA)) based on decision of a physician or a patient. Initiate administration of trastuzumab after completion of chemotherapy as a sequential combination. However, concomitant administration is allowed when combining trastuzumab with PTX, DTX and CMF. In cases of TCb (CBDCA), trastuzumab is used concomitant administration.
  Interventions: Drug: trastuzumab monotherapy; Drug: trastuzumab and chemotherapy

INTERVENTIONS:
Drug: trastuzumab monotherapy
  Other Names: Herceptin
Drug: trastuzumab and chemotherapy
  Other Names: PTX; DTX; TC; AC; EC; FEC; CMF; TCb (CBDCA)
  Arms: trastuzumab and chemotherapy

SUMMARY:
To investigate clinical positioning between trastuzumab (Herceptin) monotherapy (H group) and combination therapy of trastuzumab and chemotherapy (H+CT group) based on a randomized controlled trial in women over 70 years with human epidermal growth factor receptor type-2 (HER2) positive primary breast cancer.

DETAILED DESCRIPTION:
This study is a randomized, comparative trial of postoperative adjuvant therapies in women with HER2 (human epidermal growth factor receptor type-2)-positive primary breast cancer who are ≥70 years of age that will compare trastuzumab (Herceptin®) monotherapy (H group) and trastuzumab in combination with chemotherapy (H+CT group).

The objectives of this study are as follows.

1. To verify the clinical positioning of trastuzumab monotherapy and combined trastuzumab and chemotherapy as postoperative adjuvant therapies for the treatment of HER2-positive primary breast cancer patients who are ≥70 years of age.
2. To evaluate the safety of trastuzumab monotherapy and combined trastuzumab and chemotherapy in patients who are ≥70 years of age. In particular, to evaluate cardiac disorders that are a characteristic adverse drug reaction of trastuzumab as well as geriatric-related concerns including lipid metabolism, cerebral infarction and cognitive disorders.
3. To evaluate overall survival in patients who are ≥70 years of age using trastuzumab monotherapy or combined trastuzumab and chemotherapy.
4. To evaluate health-related quality of life (HRQOL), cost-effectiveness (utility), and conduct a comprehensive geriatric assessment (CGA) in patients who are ≥70 years of age and using trastuzumab monotherapy or combined trastuzumab and chemotherapy.
5. To establish and expand information networks by the participation of practitioners in clinical trials that are involved in general clinical practice and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed as invasive breast cancer and received curative operation for primary breast cancer.
2. Stage: 1 (tumor size [pT] > 0.5 cm), 2A, 2B or 3A/ M0
3. Female between 70 and 80 years old
4. Primary region is HER 2 positive: either 3+ overexpression by IHC or positive by FISH
5. Baseline left ventricular ejection fraction (LVEF) is ≥55% measured by echocardiography or MUGA scan within 4 weeks before registration.
6. PS: 0-1 (ECOG)
7. Sufficient organ function meeting following criteria within 4 weeks before registration:

   * Leukocyte ≥2500 mm3
   * Neutrophil ≥1500 mm3
   * Platelet ≥100 000 mm3
   * Serum total bilirubin ≤2.0 x upper limit of normal (ULN)
   * ALT (GPT) or AST (GOT) ≤2.5 x ULN
   * Serum creatinine ≤2.0 x ULN
   * ALP ≤2.5 x ULN
8. No previous endocrine therapy or chemotherapy for breast cancer
9. Signed written informed consent

Exclusion Criteria:

1. Active multiple primary cancer (synchronous multiple primary cancer and invasive cancer of other organs)
2. Postoperative histological axillary lymph node metastasis ≥4
3. Axillary lymph node is not histologically evaluated
4. Histologically confirmed positive margin in breast conservation surgery (evaluation of margin status is based on policy of site)
5. History of drug-related allergy which could hinder planned treatment
6. Any history or complication of following cardiac disorders

   * History of congestive heart failure, cardiac infarction
   * Complication requires treatment such as: ischemic cardiac disorder, arrhythmia, valvular heart disease
7. Poorly controlled hypertension (ex. Systolic arterial pressure ≥180 mmHg or diastolic blood pressure ≥100 mmHg)
8. Poorly controlled diabetes
9. Continuous visit to a medial institution is considered difficult due to deterioration of activity of daily living (ADL)
10. Difficult to participate in the trial because of psychiatric disorder or psychiatric symptoms
11. Ineligible to the trial based on decision of an investigator

Ages: 70 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 275 (Actual)
Dates: Start 2009-10-28 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Disease free survival | Patients are followed up for 8 years after initial enrollment (from Oct. 2009 through Oct. 2017).
  Disease-free survival is defined as the interval from the date of enrollment to the date of any of the following events.
  1. Local recurrence, distant metastasis
  2. Metachronous breast cancer, secondary cancer
  3. Death

SECONDARY OUTCOMES:
Overall survival | Patients are followed up for 8 years after initial enrollment (from Oct. 2009 through Oct. 2017).
  Overall survival is defined as the interval from the date of enrollment to the date of death from any cause.
Relapse-free survival | Patients are followed up for 8 years after initial enrollment (from Oct. 2009 through Oct. 2017).
  Relapse-free survival is defined as the interval from the date of enrollment to the date of any of the following events.
  1. Local recurrence, distant metastasis
  2. Death
Percentage of participants with adverse events as a measure of safety | Evaluations are performed at the time of starting the specified treatment and 2, 6, and 9 month, 1 year, 1 year 6 months, 2 years, 2 years 6 months, and 3 years after the start of treatment. Subsequently, evaluations are done at 1-year intervals.
  The following variables are evaluated: left ventricular ejection fraction, white-cell count, neutrophil count, platelet count, bilirubin level, alanine aminotransferase level, aspartate aminotransferase level, alkaline phosphatase level, and creatinine level.
Health-related QOL (HRQOL) | Evaluations are performed at the time of starting the specified treatment and 2 months, 1 year, and 3 years after the start of treatment.
  The following QOL questionnaire forms (in Japanese) are used for evaluations: FACT-G, HADS, EQ-5D, and PNQ.
Cost effectiveness analysis | Data on direct medical costs for the 3-year period after the start of the treatment are obtained from CRF. Data on direct nonmedical costs and indirect costs are obtained from questionnaires 2, 12, and 36 months after starting the treatment.
  Survey items are as follows.
  1. Direct medical costs: medical costs associated with therapy, the management of adverse events, etc.
  2. Direct nonmedical costs: transportation expenses required for medical examinations, costs of health foods, etc.
  3. Indirect costs: work-loss costs associated with treatment that are incurred directly by the patient and by their caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Sawaki, Principal Investigator — Department of Breast Oncology, Aichi Cancer Center Hospital
Locations (1):
- Aichi Cancer Center Hospital, Nagoya, Aichi-ken, Japan

REFERENCES:
- [Derived] Nozawa K, Sawaki M, Uemura Y, Tsuneizumi M, Takano T, Gondo N, Hara F, Harao M, Toyama T, Taira N, Vivancos A, Perou CM, Sanfeliu E, Braso-Maristany F, Parker JS, Buckingham W, Pare L, Villacampa G, Marin-Aguilera M, Villagrasa P, Prat A, Iwata H. HER2DX in older patients with HER2-positive early breast cancer: extended follow-up from the RESPECT trial of trastuzumab +/- chemotherapy. Nat Commun. 2025 Nov 4;16(1):9585. doi: 10.1038/s41467-025-65599-x. PMID 41188218
- [Derived] Hagiwara Y, Sawaki M, Uemura Y, Kawahara T, Shimozuma K, Ohashi Y, Takahashi M, Saito T, Baba S, Kobayashi K, Mukai H, Taira N. Impact of chemotherapy on cognitive functioning in older patients with HER2-positive breast cancer: a sub-study in the RESPECT trial. Breast Cancer Res Treat. 2021 Aug;188(3):675-683. doi: 10.1007/s10549-021-06253-0. Epub 2021 Jun 2. PMID 34080094
- [Derived] Taira N, Sawaki M, Uemura Y, Saito T, Baba S, Kobayashi K, Kawashima H, Tsuneizumi M, Sagawa N, Bando H, Takahashi M, Yamaguchi M, Takashima T, Nakayama T, Kashiwaba M, Mizuno T, Yamamoto Y, Iwata H, Ohashi Y, Mukai H, Kawahara T; RESPECT Study Group. Health-Related Quality of Life With Trastuzumab Monotherapy Versus Trastuzumab Plus Standard Chemotherapy as Adjuvant Therapy in Older Patients With HER2-Positive Breast Cancer. J Clin Oncol. 2021 Aug 1;39(22):2452-2462. doi: 10.1200/JCO.20.02751. Epub 2021 Apr 9. PMID 33835842
- [Derived] Sawaki M, Taira N, Uemura Y, Saito T, Baba S, Kobayashi K, Kawashima H, Tsuneizumi M, Sagawa N, Bando H, Takahashi M, Yamaguchi M, Takashima T, Nakayama T, Kashiwaba M, Mizuno T, Yamamoto Y, Iwata H, Kawahara T, Ohashi Y, Mukai H; RESPECT study group. Randomized Controlled Trial of Trastuzumab With or Without Chemotherapy for HER2-Positive Early Breast Cancer in Older Patients. J Clin Oncol. 2020 Nov 10;38(32):3743-3752. doi: 10.1200/JCO.20.00184. Epub 2020 Sep 16. PMID 32936713